CLINICAL TRIAL: NCT01535807
Title: CorMatrix ECM Study: To Identify Inflammatory Markers Following CABG With/Without CorMatrix's Extra Cellular Matrix (ECM)
Brief Title: CorMatrix ECM Study: To Identify Inflammatory Markers Following CABG With/Without ECM
Acronym: CorMatrix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Corvivo Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CorMatrix ECM Study
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
Keywords: Atrial Fibrillation; Cardiac surgery; Coronary Artery Bypass Graft; CorMatrix extra cellular matrix; Heart surgery; Inflammatory Biomarkers; Myocardial Infarction; identify proteomic inflammatory biomarkers
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CorMatrix Group (Active Comparator): The treatment "Cormatrix" group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  Interventions: Device: CorMatrix extra cellular matrix (ECM)
- Control (No Intervention): The control "No Intervention" group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care.

INTERVENTIONS:
Device: CorMatrix extra cellular matrix (ECM) — * Cormatrix ECM group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  * No Intervention group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care.
  Other Names: CorMatrix ECM, CorMatrix, ECM
  Arms: CorMatrix Group

SUMMARY:
The objective of this study is to identify proteomic inflammatory biomarkers to determine if there are differences in the biomarkers in patients who are treated using the CorMatrix ECM implant to close the pericardium and the patients whose pericardium is left open (the current standard of care).

DETAILED DESCRIPTION:
The pericardium's main function is to secrete proteins that ensure proper functioning within the pericardial space and to maintain pericardial pressure. Once dissected the pericardium is usually left open at the end of surgery due to the difficulty in realigning the edges and to avoid adverse effects cause by an inflammatory response. The body's inflammatory response is one of protection and healing of an injury. However many of the inflammatory biomarkers released can cause adverse outcomes after cardiac surgery, including: renal failure, myocardial infarction, atrial fibrillation, stroke and death.

CorMatrix extra cellular matrix (ECM) Technology is a Food and Drug Administration (FDA) approved unique extra cellular implant material used for pericardial closure and reconstruction. Pericardial reconstruction using porcine intestinal ECM is a novel application. ECM combines the innate attributes of nature with the precision of science to help the heart heal itself. It is an acellular biomaterial that does not encapsulate when surgically implanted, but is gradually remodeled, leaving behind organized and healthy tissue. The body's tissue begins remodeling at the surgical site while the ECM maintains the needed tissue support. When implanted, the ECM acts as a scaffold into which the patient's cells migrate and integrate, stimulating the patient's natural wound-healing mechanisms. As the patient's cells become active, they lay down their own collagen, which matures over time to form strong and permanent tissue repair without leaving behind permanent foreign material. Because the ECM contains primarily collagen, the device is gradually replaced as the patient's tissue gradually turns over in a natural state of self-renewal.

A retrospective study compared the incidence of post operative atrial fibrillation (POAF) in patients treated with the CorMatrix ECM for pericardial closure following isolated coronary artery bypass graft (CABG) versus patients not treated with the patch. The retrospective study comprised of 222 patients. 111 were treated with the CorMatrix ECM and the other 111 were not. Results showed POAF in 34 of 111 control patients but only 20 in 111 CorMatrix ECM treated patients, indicating a 54% decrease in the risk of POAF in the CorMatrix ECM treated patients. This study shows a statistically significant reduction in the risk of POAF in patients undergoing an isolated CABG with pericardial closure using the CorMatrix ECM.

This is an unblinded, randomized study to identify proteomic inflammatory biomarkers to determine if there are differences in the biomarkers in patients who are treated using the CorMatrix ECM implant to close the pericardium and the patients whose pericardium is left open (the current standard of care). The study will be located at the Inova Heart and Vascular Institute (IHVI). The CorMatrix ECM will be implanted during the CABG surgical procedure in the IHVI cardiovascular operating rooms (CVOR).

Sixty (60) patients who are routinely scheduled for a CABG will be recruited and randomly assigned to one of the two groups. There will be thirty (30) patients in each group. The control "No Intervention" group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care. The treatment "Cormatrix" group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.

Pericardial fluid and blood samples will be collected from all patients. Pericardial fluid and blood samples will undergo novel nanoparticle based biomarker discovery technology to harvest proteomic biomarkers at the George mason University. In addition, patients will have their cardiac rhythm continually assessed during their hospital stay and then at their follow up appointments with their surgeon and cardiologist to determine whether they developed POAF post discharge.

Both genders, greater than eighteen (18) years of age, will be included in the research. There are no enrollment restrictions based upon race or ethnic origin and it is expected their inclusion will be representative of the population undergoing CABG at IHVI. Pregnant women are excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Subject must be selected as a candidate for isolated Coronary Artery Bypass Graft (CABG) procedure
* Subject has a Left Ventricular Ejection Fraction (LVEF) of ≥30%
* Subject is able and willing to provide written informed consent and HIPAA authorization
* Subject has a life expectancy of at least one year

Exclusion Criteria:

* Subject is scheduled for other concomitant surgical procedures (carotid surgery included)
* Subject has a known hypersensitivity to porcine material
* Subject has a religious or cultural objection to the use of blood or porcine products
* Subject is scheduled for Off Pump Coronary Artery Bypass procedures (OPCAB)
* Subject has a history of diagnosed treated or un-treated pre-operative atrial fibrillation or any other type of cardiac arrhythmia
* Subject has a history of anti-arrhythmic drug treatment in the past six (6) months
* Subject has an implantable cardiac device (e.g., pacemakers, implantable cardioverter defibrillators)
* Subject has a history of an accessory pathway disorder (e.g., Wolff-Parkinson-White syndrome)
* Subject has a documented myocardial infarction (MI) within six (6) weeks prior to study enrollment
* Subject needs emergent cardiac surgery (i.e., cardiogenic shock)
* Subject requires intra-aortic balloon pump or intravenous inotropes
* Subject has had an infection within six (6) weeks preceding surgery requiring antibiotic therapy
* Subject is on pre-surgical immunosuppressive therapy (corticosteroids included)
* Subject has chronic inflammatory disease (leukemia, lymphoma, arthritis, rheumatoid, lupus, Crohn's disease, ulcerative colitis, hepatitis C, HIV)
* Subject has had therapeutic radiation to the pericardium, either prior to surgery or expected during the three (3) week period following surgery
* There is an inability to approximate the graft and pericardium edge along the entire extent of the defect
* Subject is incarcerated
* Subject is participating in concomitant research studies of investigational products (e.g., Appendage closure devices, septal defect patches)
* Subject is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Inova Health Systems
Locations (1):
- Inova Heart and Vascular Institute, Falls Church, Virginia, United States

REFERENCES:
- See also: ECM Technologies by CorMatrix — http://www.cormatrix.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- CorMatrix Group: The treatment "Cormatrix" group will receive the CorMatrix extra cellular matrix (ECM) during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  CorMatrix ECM: - Cormatrix ECM group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  - No Intervention group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care.
Period: Overall Study
Arm/Group | CorMatrix Group | Control
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Data collection error | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- CorMatrix Group: The treatment "Cormatrix" group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  CorMatrix extra cellular matrix (ECM): - Cormatrix ECM group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  - No Intervention group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care.
- Total: Total of all reporting groups
Arm/Group | CorMatrix Group | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.18 (9.88) | 60.17 (9.84) | 60.30 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Cytokine Levels in Participant Sera From Pre-surgery Baseline to Day 3 Post-surgery.
Description: Percentage change in Inflammatory Cytokine Levels in serum derived from participant blood sample that underwent novel nanoparticle-based biomarker harvesting technology to capture and isolate global low molecular weight (LMW) proteome. Peptides from captured proteomes are detected with reversed-phase liquid chromatography/electrospray tandem mass spectrometry (LC-MS/MS).
  Inflammatory cytokines include Interleukin 6 (IL6), Interleukin 8 (IL8), Interleukin 2 Receptor (IL2R), Tumor Necrosis Factor (TNF), and Lipopolysaccharide Binding Protein (LBP). The measure of their respective levels is defined here as the Spectral Count from LC-MS/MS analysis.
  Percentage change of Spectral Counts is the difference of Day 3 post-surgery and pre-surgical baseline relative to the pre-surgical baseline.
Time Frame: Baseline and and Post-Op day 3
Measure: Mean (Standard Error); unit: Percent Change
Groups:
- CorMatrix Group: The treatment "Cormatrix" group will receive the CorMatrix ECM (Extra Cellular Matrix) during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  CorMatrix ECM: - Cormatrix ECM group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  - No Intervention group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care.
Arm/Group | CorMatrix Group | Control
Number analyzed (Participants) | 20 | 20
Percent Change
  IL6 (Interleukin 6) | 645 (400) | 767 (380)
  IL8 (Interleukin 8) | 44 (2) | 28 (16)
  IL2R (Interleukin 2 Receptor) | 35 (29) | 31 (25)
  TNF (Tumor Necrosis Factor) | 5 (3) | 7 (5)
  LBP (Lipopolysaccharide Binding Protein) | 190 (45) | 197 (57)

2. Secondary Outcome: Occurrences of Post Operative Atrial Fibrillation (POAF)
Description: Number of patients that were determined to have Post Operative Atrial Fibrillation by electrocardiograph within 30 days of surgery
Time Frame: Up to 30 days post surgery
Measure: Count of Participants; unit: Participants
Groups:
- CorMatrix Group: The treatment "Cormatrix" group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  CorMatrix ECM: - Cormatrix ECM group will receive the CorMatrix ECM during surgery for the closure of the pericardium according to the specific recommended surgical technique.
  - No Intervention group will not receive the CorMatrix ECM during surgery, leaving the pericardium open according to current standard of care.
Arm/Group | CorMatrix Group | Control
Number analyzed (Participants) | 20 | 20
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | CorMatrix Group | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No